CLINICAL TRIAL: NCT03689478
Title: A Pilot Study on the Use of Immediate Hyperthermic Intravesical Chemotherapy Following Transurethral Resection of Bladder Tumour (I-HIVEC Study)
Brief Title: Use of Immediate Hyperthermic Intravesical Chemotherapy Following TURBT
Acronym: I-HIVEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE Ref. No. 2018.206
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer; Hyperthermia; Chemotherapy Effect
Keywords: Hyperthermic intravesical chemotherapy; Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Prospective single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperthermic intravesical chemotherapy (Experimental): Intravesical instillation of 40mg mitomycin C at 43 degrees for 60 minutes immediately after transurethral resection of bladder tumour
  Interventions: Other: Hyperthermic intravesical chemotherapy

INTERVENTIONS:
Other: Hyperthermic intravesical chemotherapy — Intravesical instillation of 40mg mitomycin C at 43 degrees for 60 minutes immediately after transurethral resection of bladder tumour

SUMMARY:
This is a prospective single-arm pilot study investigating the safety and feasibility of giving hyperthermic intravesical chemotherapy immediately following transurethral resection of bladder tumour.

DETAILED DESCRIPTION:
The Combat Bladder Recirculation System (BRS) is a CE marked device which has been used in over 200 sites in Europe. It is an aluminum heat exchanger that allows hyperthermic intravesical chemotherapy (HIVEC) at 43±0.2 degrees for patients with bladder cancer. Previous studies showed that the Combat BRS could warm the entire bladder wall to the target temperature with excellent safety parameters. The flow rates and pressure levels are kept low during the HIVEC treatment. A previous study has demonstrated the safety and tolerability of HIVEC as a maintenance therapy for patients with non-muscle-invasive bladder cancer (NMIBC), and two randomized controlled trials are underway to demonstrate its efficacy in terms of disease recurrence and progression. On the other hand, the use of HIVEC immediately following transurethral resection of bladder tumour (TURBT) remains largely unexplored. It is the investigators' current practice to give intravesical mitomycin C (MMC) to all patients who have endoscopically NMIBC with complete resection, provided that there are no bladder perforations being noted. In this study, the investigators shall evaluate the safety and feasibility of hyperthermia in addition to the current practice of intravesical MMC alone immediately following TURBT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above with informed consent

Exclusion Criteria:

* ECOG performance status ≥2
* ASA 4 or above
* History of bleeding disorder
* Any use of anti-coagulants
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
30-day complications | Thirty days after the experimental treatment
  Complications which occur within 30 days after the experimental treatment

SECONDARY OUTCOMES:
Hyperthermic intravesical chemotherapy instillation rate | One day after surgery
  Rate of hyperthermic intravesical chemotherapy instillation given after the operation
Duration of urethral catheterisation | Two days after the experimental treatment
  Duration of urethral catheterisation after the experimental treatment
Rate of bladder irrigation | One day after the experimental treatment
  Rate of bladder irrigation given after the experimental treatment
Duration of bladder irrigation | Two days after the experimental treatment
  Duration of bladder irrigation after the experimental treatment
Hospital stay | Three days after the experimental treatment
  Duration of hospital stay for the experimental treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Schooneveldt G, Bakker A, Balidemaj E, Chopra R, Crezee J, Geijsen ED, Hartmann J, Hulshof MC, Kok HP, Paulides MM, Sousa-Escandon A, Stauffer PR, Maccarini PF. Thermal dosimetry for bladder hyperthermia treatment. An overview. Int J Hyperthermia. 2016 Jun;32(4):417-33. doi: 10.3109/02656736.2016.1156170. Epub 2016 May 1. PMID 27132465
- [Background] Owusu RA, Abern MR, Inman BA. Hyperthermia as adjunct to intravesical chemotherapy for bladder cancer. Biomed Res Int. 2013;2013:262313. doi: 10.1155/2013/262313. Epub 2013 Sep 1. PMID 24073396
- [Background] Kok HP, Wust P, Stauffer PR, Bardati F, van Rhoon GC, Crezee J. Current state of the art of regional hyperthermia treatment planning: a review. Radiat Oncol. 2015 Sep 17;10:196. doi: 10.1186/s13014-015-0503-8. PMID 26383087
- [Background] Teicher BA, Kowal CD, Kennedy KA, Sartorelli AC. Enhancement by hyperthermia of the in vitro cytotoxicity of mitomycin C toward hypoxic tumor cells. Cancer Res. 1981 Mar;41(3):1096-9. PMID 7459853